CLINICAL TRIAL: NCT04498039
Title: Reducing Symptoms of Multiple Sclerosis Using Non-invasive Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: H2008-0252
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study is a within-subject blinded randomized control design. Twenty chronic MS subjects with an identified gait disturbance were assigned to either an active or control group. Both groups completed a 14-week intervention program using a standardized combination of exercise and a device that provided electrical stimulation to the tongue. Those in the active group received electrical stimulation on the tongue that they could perceive.
  Those in the control group used a device that did not provide a physiologically significant stimulus and was not perceivable. Subjects were assessed with the Dynamic Gait Index (DGI).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Electrical stimulation to the tongue is delivered via the Portable Neuromodulation Stimulator (PoNS™) device . The PoNS™ device is held in place lightly by the lips and teeth around a rectangular tab that goes into the mouth and rests on the anterior, superior part of the tongue. Active subjects will be able to feel the sensation.
  Interventions: Device: Portable Neuromodulation Stimulator
- Control (Sham Comparator): Electrical stimulation to the tongue will be delivered via the Portable Neuromodulation Stimulator (PoNS™) device . The PoNS™ device is held in place lightly by the lips and teeth around a rectangular tab that goes into the mouth and rests on the anterior, superior part of the tongue. Control subjects will be informed that while they may not feel the electrotactile stimulation, they are in-fact receiving a low level signal.
  Interventions: Device: Portable Neuromodulation Stimulator

INTERVENTIONS:
Device: Portable Neuromodulation Stimulator — Examining the effect of targeted physical therapy with and without cranial nerve non-invasive neuromodulation (CN-NINM), on the walking ability of people with MS who exhibit a dysfunctional gait. Adopting a rehabilitative strategy using neuromodulation of the cranial nerves via electrical stimulation of the tongue to enhance the plasticity of the brain.
  Other Names: PoNS

SUMMARY:
This study sought to examine the effect of targeted physical therapy with and without cranial nerve non-invasive neuromodulation (CN-NINM), on the walking ability of people with MS who exhibited a dysfunctional gait.

DETAILED DESCRIPTION:
Background: This study sought to examine the effect of targeted physical therapy with and without cranial nerve non-invasive neuromodulation (CN-NINM), on the walking ability of people with MS who exhibited a dysfunctional gait. The investigators hypothesized that subjects who received electrical stimulation would have greater improvement than those who had a control device after a 14-week intervention. Gait disturbance is a common problem for people with multiple sclerosis (MS). The investigators have developed an effective rehabilitative strategy using neuromodulation of the cranial nerves via electrical stimulation of the tongue to enhance the plasticity of the brain.

Methods: The study is a within-subject blinded randomized control design. Twenty chronic MS subjects with an identified gait disturbance were assigned to either an active or control group. Both groups completed a 14-week intervention program using a standardized combination of exercise and a device that provided electrical stimulation to the tongue. Those in the active group received electrical stimulation on the tongue that they could perceive. Those in the control group used a device that did not provide a physiologically significant stimulus and was not perceivable. Subjects were assessed with the Dynamic Gait Index (DGI).

ELIGIBILITY:
All subjects are initially evaluated for inclusion/exclusion on the Kurtzke Expanded Disability Status Scale (EDSS), a test typically administered by their healthcare provider as an ongoing part of standard therapy for M.S

Inclusion Criteria:

* Relapsing remitting MS ("RRMS"), primary progressive MS ("PPMS"), or secondary progressive MS ("SPMS") without relapse within 6 months of enrollment;
* EDSS score of 3.0 - 6.0 ;
* No changes in medication within 3 months of enrollment;
* Ability to walk 20 minutes on a treadmill (with handrail support as needed) without rest;
* Provided informed consent and willing to participate.

Exclusion Criteria:

• Major co-morbidities, especially other neurological disorders, uncontrolled pain, hypertension, diabetes, or oral health problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index DGI | 14 weeks
  The Dynamic Gait Index (DGI) is a clinician-scored index of 8 gait tasks which was developed as a clinical tool for assessing gait, balance, and fall risk by evaluating dynamic balance. Tasks include steady state walking, changing speeds while walking, walking with horizontal and vertical head turns, walking around and stepping over objects, walking to a pivot turn and stop, and traversing stairs. The maximum total individual score is 24 points (0-3 on each task), with higher scores indicating better function. A 4-point change in DGI would require an improvement of at least one level on four of 8 tasks, or multiple levels of improvement on several tasks. Thus, a 4-point change represents a clinically significant difference that is generally measurable without excessive variability.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E Tyler, P.E, M.S, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No